CLINICAL TRIAL: NCT03709147
Title: Exploiting Metformin Plus/Minus Cyclic Fasting Mimicking Diet (FMD) to Improve the Efficacy of First Line Chemo-immunotherapy in Advanced LKB1-inactive Lung Adenocarcinoma
Brief Title: Metformin Plus/Minus Fasting Mimicking Diet to Target the Metabolic Vulnerabilities of LKB1-inactive Lung Adenocarcinoma
Acronym: FAME
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marina Garassino (Other)
Responsible Party: Sponsor-Investigator, Marina Garassino, Principal Investigator; Head of Unit of Thoracic Oncology, Medical Oncology Department, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Organization: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT 45/18
Record Dates: First submitted 2018-09-20; First posted 2018-10-17 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Advanced LKB1-inactive Lung Adenocarcinoma
Keywords: LKB1-inactive adenocarcinoma; Cisplatin-pemetrexed; Metformin; Fasting-mimicking diet (FMD); Progression-free survival
MeSH Terms: interventions — Metformin; Cisplatin; Carboplatin; Pemetrexed; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Single Institution, open-labeled, triple arm, non-comparative phase II trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- FAME arm (Experimental): * cisplatin 75 mg/mq every three weeks OR carboplatin (CBDCA) at an area under the curve (AUC) of 5 every three weeks, up to a maximum of 4 cycles
  * pemetrexed 500 mg/mq every three weeks
  * pembrolizumab 200 mg flat dose every three weeks
  * metformin hydrochloride up to a daily dosage of 1500 mg
  * every-three week, 5-day Fasting-mimicking diet (FMD), up to a maximum of 4 cycles
  Interventions: Drug: Metformin Hydrochloride; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Dietary Supplement: Fasting-mimicking diet; Drug: Pembrolizumab
- MERCY arm (Experimental): * cisplatin 75 mg/mq every three weeks OR carboplatin (CBDCA) at an area under the curve (AUC) of 5 every three weeks, up to a maximum of 4 cycles
  * pemetrexed 500 mg/mq every three weeks
  * pembrolizumab 200 mg flat dose every three weeks
  * metformin hydrochloride up to a daily dosage of 1500 mg
  Interventions: Drug: Metformin Hydrochloride; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Drug: Pembrolizumab
- BORN arm (No Intervention): Standard clinical approach.

INTERVENTIONS:
Drug: Metformin Hydrochloride — Metformin 1500 mg/day up to disease progression or unacceptable toxicity Every-21-days, 5-day Fasting-mimicking diet (FMD)
  Other Names: Metformin
  Arms: FAME arm; MERCY arm
Drug: Cisplatin — Intravenous cisplatin, administered at a dosage of 75 mg/mq every three weeks for a maximim of 4 consecutive cycles
  Other Names: CDDP
  Arms: FAME arm; MERCY arm
Drug: Carboplatin — Carboplatin at an area-under-the-curve (AUC) of 5, administered intravenously every-three weeks for a maximum of 4 consecutive cycles
  Other Names: CBDCA
  Arms: FAME arm; MERCY arm
Drug: Pemetrexed — Pemetrexed, administered intravenously at the dose of 500 mg/mq every-three weeks up to a maximum of 4 cycles in combination with platinum compounds, and then as a maintenance treatments in patients not undergoing disease progression after the first 4 chemotherapy cycles
  Arms: FAME arm; MERCY arm
Dietary Supplement: Fasting-mimicking diet — 5-day fasting-mimicking diet regimen, consisting of 700 KCal on day 1, 300 KCal on days 2-4, and 450 KCal on day 5, to be repeated every three weeks up to a maximum of 4 cycles
  Other Names: FMD
  Arms: FAME arm
Drug: Pembrolizumab — Pembrolizumab, administered intravenously at the flat dose of 200 mg every-three weeks up to a maximum of 4 cycles in combination with platinum compounds, and then as a maintenance treatments in patients not undergoing disease progression after the first 4 chemotherapy cycles
  Arms: FAME arm; MERCY arm

SUMMARY:
Lung adenocarcinoma with inactive LKB1 has emerged as a particularly aggressive form of lung cancer, with poor response to immune checkpoint inhibitors. Recent preclinical evidences have demonstrated that LKB1-inactive lung adenocarcinoma is characterized by specific metabolic vulnerabilities, which make it hypersensitive to energetic crisis. For instance, by inhibiting mitochondrial metabolism and reducing ATP availability to cancer cells, the antidiabetic compound metformin has anticancer activity and prevents acquired resistance to cisplatin in lung adenocarcinoma with inactive LKB1. Similarly to metformin, glucose starvation, which can be recapitulated in vivo by cyclic fasting or fasting-mimicking diet (FMD), can cause metabolic crisis in these neoplasms. In this trial, the investigators will assess for the first time the efficacy of combining standard-of-care platinum-based chemoimmunotherapy with metformin plus/minus FMD in patients with LKB1-inactive, advanced lung adenocarcinoma.

DETAILED DESCRIPTION:
Lung cancer is one of the most common malignancies and tumor-related causes of death worldwide. In the last years, significant advances have been observed in the treatment of non small cell lung cancer, in particular for the population of patients with a driver genetic mutation like EGFR and ALK. For the remaining cases, the main novelty has been represented by immunotherapy with anti-PD1/PDL1 agents, which have proved a benefit over previous standard of care (platinum-based chemotherapy in first line and docetaxel in second line). , Only patients wih tumors expressing high PD-L1 levels have had access to immunotherapy alone as first line treatment. For all the remaining cases, the standard-of-care treatment in the first-line setting has remained platinum-based chemotherapy for several years. This algorithm has been recently changed by the approval of combined chemotherapy(platinum salt + pemetrexed) and immunotherapy (pembrolizumab) as a first-line therapy for patients with lung adenocarcinoma and low/absent PD-L1 expression. This regimen has entered into clinical practice following the positive results of a clinical trial, showing superior outcome with the combination than with chemotherapy alone. Lung adenocarcinoma with LKB1 mutations or macro/micro deletions has a particularly aggressive behavior and seems to be resistant to the effects of immunotherapy, either alone or in combination with chemotherapy. Indeed, such a population appears to be disadvantaged as regards therapeutic options and requires the development of different approaches. LKB1 enzyme is involved in intracellular pathways that are crucial in the regulation of cancer cell metabolism. Metabolic reprogramming is a key step in tumorigenesis and several metabolic pathways, including glucose uptake and utilization, or lipid biosynthesis and utilization, are deregulated in cancer cells compared to their normal counterpart. Cells with hypo-active or inactive LKB1 are peculiar in that they show an exquisite vulnerability to energetic deprivation. Indeed, they are unable to survive when exposed to nutrient deprivation or drugs that affect cancer cell bioenergetics or specific metabolic processes. In particular, the class of drugs known as biguanides, which include the antidiabetic compound metformin, are able to inhibit mitochondrial metabolism and to reduce the intracellular concentration of ATP, and have shown antitumor activity in mouse xenografts of LKB1-mutated lung adenocarcinomas. Based on the well known effects of metformin on cancer cell metabolism, as well as on preclinical evidence showing synergistic activity of cisplatin and metformin in lung cancer cell lines and animal models with LKB1 deletion, we hypothesize that combining chemoimmunotherapy (platinum salt + pemetrexed + pembrolizumab) with either metformin (MERCY arm), or metformin plus a lowcalorie, low-carbohydrate, low-protein diet also known as Fasting Mimicking Diet (FMD) (FAME arm), may improve the efficacy of standard treatment alone for patients with LKB1-inactive lung adenocarcinoma.

The patients considered eligible and enrolled in the study will be included in FAME, MERCY or BORN arms according to the aforementioned eligibility criteria. Patients in each arm will receive the following treatment:

* FAME -> up to a maximum of 4 cycles of a platinum salt + pemetrexed + pembrolizumab in association to metformin and to tri-weekly, 5 day-long cycles of FMD.
* MERCY -> up to a maximum of 4 cycles of a platinum salt + pemetrexed + pembrolizumab in association to metformin.
* BORN -> standard treatment at investigator's choice or observation only in case of clinical conditions contraindicating any active therapy.

In both arms FAME and MERCY, the patients with stable or responding disease after 4 cycles of chemotherapy will continue with maintenance pemetrexed and pembrolizumab in association to metformin until disease progression and/or inacceptable toxicity.

ELIGIBILITY:
FAME arm (chemo-immunotherapy + metformin + FMD):

Inclusion criteria:

1. Age included between 18 and 75 years.
2. Histologically confirmed diagnosis of LKB1-inactive lung adenocarcinoma, as defined on the basis of absence of LKB1 expression at immunoistochemistry, and/or presence of pathogenic LKB1 mutations/deletions at next-generation sequencing analysis.
3. Absence of EGFR mutations, ALK and ROS-1 rearrangements, and absence of high expression of PD-L1 (≥ 50% in immunohistochemistry).
4. Advanced disease, defined as unresectable, locally advanced (stage IIIB) or metastatic (stage IV) lung adenocarcinoma, which is not candidate to be treated with concomitant or sequential definitive chemo-radiation.
5. Signed and dated informed consent, indicating that the patient has been informed on all the aspects of the study prior to the enrollment.
6. Patient's will able to respect the protocol recommendations about the FMD regimen, as well as about laboratory tests and other procedures.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
8. In case of presence of brain metastases, the patient can be candidated to be enrolled in the study, provided that neurologic symptoms are absent, the patient does not need radiotherapy or treatment with steroids at a dose ≥ 4 mg per day of dexamethasone or analogues.
9. Adequate bone marrow and organ function, defined as follows:

   * absolute neutrophil count ≥ 1.5 x 103/L;
   * platelet count ≥ 100 x 103/L;
   * hemoglobin ≥ 9.0 g/dL;
   * serum albumin-corrected calcium within normal range or with anomalies graded ≤ 1 according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 if not clinically significant;
   * potassium within normal range or corrected with supplements;
   * glomerular filtration rate (GFR) > 60 mL/min, estimated on a 24-hour urine exam and calculated from serum creatinine with Cockroft-Gault formula;
   * uric acid < 10 mg/dL;
   * AST and ALT ≤ 2.5 times upper normal limits, or ≤ 5 times upper normal limits in case of liver metastases;
   * serum bilirubin < 1.5 times upper normal limits, except for patients with Gilbert syndrome who will be considered amenable to be enrolled if total bilirubin is < 3.0 times upper normal limits or direct bilirubin is < 1.5 times upper normal limits;
   * serum albumin > 3 g/dL.
10. Fasting plasma glucose concentration ≤ 200 mg/dL.
11. For women of childbearing potential, consent to maintain abstinence from sexual intercourse or to use highly effective contraceptive methods (that is, with a failure rate < 1% per year) for the whole duration of the study and for almost 30 days after the conclusion of the FMD. Abstinence is acceptable only if in line with the patient's lifestyle. Adequate contraceptive methods include tube ligation, male sterilization, hormone implants, injectable or oral hormone contraceptives and some intra-uterine devices. Alternatively, two different contraceptive methods must be combined (e.g. two barrier methods like condom and cervical cap) in order to obtain a failure rate <1% per year. Barrier methods must always be associated to a sperm killer.

Exclusion criteria:

1. Previous systemic therapies for advanced lung cancer.
2. Evidence of disease relapse within 6 months from the conclusion of adjuvant or neoadjuvant platinum-based chemotherapy.
3. Diagnosis of other malignancies in the previous 5 years, except for adequately treated basal or squamous skin cancer or radically excised cervical cancers. Other malignancies diagnosed more than 5 years before the diagnosis of lung cancer must have been radically treated without evidence of relapse at the time of patient enrollment.
4. Body mass index (BMI) < 20 kg/m2.
5. Anamnesis of alcohol abuse.
6. Non-intentional weight loss ≥ 5% in the previous 3 months, unless the patient has a BMI > 25 kg/ m2 at the time of enrollment in the study, or non-intentional weight loss of ≥ 10% in the previous 3 months, unless the patients has a BMI > 22 kg/m2 at the time of the enrollment in the study. In both cases, weight must have remained stable for at least one month.
7. Active pregnancy or breast feeding.
8. Active B or C hepatitis.
9. Serious infection in the previous 4 weeks before the start of FMD, including, but not limited to, potential hospitalizations for complications of infections, bacteriemia or serious pneumonitis.
10. Active autoimmune diseases requiring systemic treatments (e.g. systemic steroids or immune suppressants).
11. Recent diagnosis of hypothyroidism requiring systemic substitutive hormonal therapy and without stabilization of hormonal profile (fT3, fT4 and TSH within the normal range).
12. Diagnosis of type 1 or 2 diabetes mellitus requiring pharmacologic therapy (including, but not limited to, insulin, secretagogues and metformin).
13. Serious impairment of gastrointestinal function or gastrointestinal disease potentially altering nutrient digestion or absorption during re-alimentation phase (e.g. active gastric or intestinal ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small intestine resection).
14. Anamnesis of human immunodeficiency virus (HIV).
15. Anamnesis of clinically significant heart disease including:

    1. angina pectoris, coronary bypass, symptomatic pericarditis, myocardial infarction in the previous 12 months from the beginning of experimental therapy;
    2. congestive heart failure (NYHA III-IV).
16. Anamnesis of cardiac arrhythmias (e.g. ventricular tachycardia, chronic atrial fibrillation, complete bundle branch block, high grade atrio-ventricular block like bi-fascicular block, type II Mobitz and third grade atrio-ventricular block, nodal arrhythmias, supra-ventricular arrhythmias) or conduction abnormalities in the previous 12 months from the beginning of experimental therapy.
17. Reduction in left ventricular ejection fraction to < 50% at the cardiac scan with radionuclides or at echocardiography.
18. Previous episodes of symptomatic hypotension leading to loss of consciousness.
19. Plasma fasting glucose ≤ 65 mg/dL.
20. Active therapy with systemic steroids at a dose ≥ 25 mg per day of prednisone or equivalent for any reason.
21. Medical or psychiatric comorbidities rendering the patient not candidate to the clinical trial, according to the investigator's judgement.
22. pO2 < 60 mmHg, lactates above normal limits and pH value below normal limits at arterial hemogasanalysis.
23. Need for chronic oxygen therapy.
24. Other cardiac, liver, lung or renal comorbidities, not specified in the previous inclusion or exclusion criteria, but potentially exposing the patient to a high risk of lactic acidosis.

MERCY arm (chemo-immunotherapy + metformin):

Inclusion criteria:

1. Age ≥18 years.
2. Histologically confirmed diagnosis of LKB1-inactive lung adenocarcinoma, as defined on the basis of absence of LKB1 expression at immunoistochemistry, and/or presence of pathogenic LKB1 mutations/deletions at next-generation sequencing analysis.
3. Absence of EGFR mutations, ALK and ROS-1 rearrangements, and absence of high expression of PD-L1 (≥ 50% in immunohistochemistry).
4. Advanced disease, defined as unresectable, locally advanced (stage IIIB) or metastatic (stage IV) lung adenocarcinoma, which is not candidate to be treated with concomitant or sequential definitive chemo-radiation.
5. Signed and dated informed consent, indicating that the patient has been informed on all the aspects of the study prior to the enrollment.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
7. Adequate bone marrow and organ function, defined as follows:

   * absolute neutrophil count ≥ 1.5 x 103/L;
   * platelet count ≥ 100 x 103/L;- hemoglobin ≥ 9.0 g/dL;
   * serum albumin-corrected calcium within normal range or with anomalies graded ≤ 1 according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 if not clinically significant;
   * potassium within normal range or corrected with supplements;
   * glomerular filtration rate (GFR) > 60 mL/min, estimated on a 24-hour urine exam and calculated from serum creatinine with Cockroft-Gault formula;
   * uric acid < 10 mg/dL;
   * AST and ALT ≤ 2.5 times upper normal limits, or ≤ 5 times upper normal limits in case of liver metastases;
   * serum bilirubin < 1.5 times upper normal limits, except for patients with Gilbert syndrome who will be considered amenable to be enrolled if total bilirubin is < 3.0 times upper normal limits or direct bilirubin is < 1.5 times upper normal limits;
   * serum albumin > 3 g/dL.
8. For women of childbearing potential, consent to maintain abstinence from sexual intercourse or to use highly effective contraceptive methods (that is, with a failure rate < 1% per year) for the whole duration of the study and for almost 30 days after the conclusion of the metformin treatment. Abstinence is acceptable only if in line with the patient's lifestyle. Adequate contraceptive methods include tube ligation, male sterilization, hormone implants, injectable or oral hormone contraceptives and some intra-uterine devices. Alternatively, two different contraceptive methods must be combined (e.g. two barrier methods like condom and cervical cap) in order to obtain a failure rate <1% per year. Barrier methods must always be associated to a sperm killer.

Exclusion criteria:

1. Previous systemic therapies for advanced lung cancer.
2. Evidence of disease relapse within 6 months from the conclusion of adjuvant or neoadjuvant platinum-based chemotherapy.
3. Diagnosis of other malignancies in the previous 5 years, except for adequately treated basal or squamous skin cancer or radically excised cervical cancers. Other malignancies diagnosed more than 5 years before the diagnosis of lung cancer must have been radically treated without evidence of relapse.
4. Anamnesis of alcohol abuse.
5. Active pregnancy or breast feeding.
6. Active B or C hepatitis.
7. Serious infection in the previous 4 weeks before the start of metformin treatment, including, but not limited to, potential hospitalizations for complications of infections, bacteriemia or serious pneumonitis.
8. Active autoimmune diseases requiring systemic treatments (e.g. systemic steroids or immune suppressants).
9. Recent diagnosis of hypothyroidism requiring systemic substitutive hormonal therapy and without stabilization of hormonal profile (fT3, fT4 and TSH within the normal range).
10. Diagnosis of type 1 or 2 diabetes mellitus requiring pharmacologic therapy (including, but not limited to, insulin, secretagogues and metformin).
11. Serious impairment of gastrointestinal function or gastrointestinal disease potentially altering nutrient digestion or absorption during re-alimentation phase (e.g. active gastric or intestinal ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small intestine resection).
12. Anamnesis of human immunodeficiency virus (HIV).
13. Anamnesis of clinically significant heart disease including:

    1. angina pectoris, coronary bypass, symptomatic pericarditis, myocardial infarction in the previous 12 months from the beginning of experimental therapy;
    2. congestive heart failure (NYHA III-IV).
14. Anamnesis of cardiac arrhythmias (e.g. ventricular tachycardia, chronic atrial fibrillation, complete bundle branch block, high grade atrio-ventricular block like bi-fascicular block, type II Mobitz and third grade atrio-ventricular block, nodal arrhythmias, supra-ventricular arrhythmias) or conduction abnormalities in the previous 12 months from the beginning of experimental therapy.
15. Reduction in left ventricular ejection fraction to < 50% at the cardiac scan with radionuclides or at echocardiography.
16. Medical or psychiatric comorbidities rendering the patient not candidate to the clinical trial, according to the investigator's judgement.
17. pO2 < 60 mmHg, lactates above normal limits and pH value below normal limits at arterial hemogasanalysis.
18. Need for chronic oxygen therapy.
19. Other cardiac, liver, lung or renal comorbidities, not specified in the previous inclusion or exclusion criteria, but potentially exposing the patient to a high risk of lactic acidosis.

BORN (observational arm):

Inclusion criteria:

1. Age ≥18 years.
2. Histologically confirmed diagnosis of LKB1-inactive lung adenocarcinoma, as defined on the basis of absence of LKB1 expression at immunoistochemistry, and/or presence of pathogenic LKB1 mutation at next-generation sequencing analysis.
3. Absence of EGFR mutations, ALK and ROS-1 rearrangements, and absence of high expression of PD-L1 (≥ 50% in immunohistochemistry).
4. Advanced disease, defined as unresectable, locally advanced (stage IIIB) or metastatic (stage IV) lung adenocarcinoma, which is not candidate to be treated with concomitant or sequential definitive chemo-radiation.
5. Signed and dated informed consent, indicating that the patient has been informed on all the aspects of the study prior to the enrollment.
6. At least one exclusion criteria of FAME and MERCY arm.

Exclusion criteria:

None

Patients who are eligible for the FAME arm will be preferentially proposed to be enrolled in the FAME. If they refuse, then they will be proposed to be enrolled in the MERCY arm. If they also refuse to be enrolled in the MERCY arm, they will be proposed to be enrolled in the BORN arm.

Patients who are eligible for the MERCY arm will be preferentially proposed to be enrolled in the MERCY arm; if they refuse, the will be proposed to be enrolled in the BORN arm.

Finally, patients who are ineligible for both the FAME and MERCY arms will be proposed to be enrolled in the BORN arm.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2018-10-30 (Actual); Primary Completion 2023-09-10 (Estimated); Study Completion 2023-09-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 60 months
  Progression-free survival (PFS), as defined as the time between treatment initiation and disease progression or patient death from any cause, whichever came first

SECONDARY OUTCOMES:
Grade 3/4 adverse events (AEs) | 60 months
  Incidence (%) Grade 3/4 adverse events (AEs)
Treatment-related adverse events | 60 months
  Incidence (%) of treatment-related adverse events
Patient compliance to the experimental treatment | 40 months
  Patient compliance to the experimental treatment, as evaluated from the analysis of daily food diaries
Objective response rate (ORR) | 40 months
  Objective response rate (ORR), as measured with Radiologic Evaluation Criteria In Solid Tumors (RECIST) version 1.1.
Overall survival (OS) | 60 months
  Overall survival (OS), as defined as the time between treatment initiation and patient death from any cause
Effect of the experimental treatment on plasma glucose levels | 40 months
  Effect of the experimental treatment on plasma glucose levels
Effect of the experimental treatment on serum insulin levels | 40 months
  Effect of the experimental treatment on serum insulin levels
Effect of the experimental treatment on serum IGF-1 levels | 40 months
  Effect of the experimental treatment on serum IGF-1 levels
Effect of the experimental treatment on plasma fatty acids | 40 months
  Effect of the experimental treatment on plasma fatty acids, measured through mass spectrometry analysis
Effect of the experimental treatment on urinary ketones | 40 months
  Effect of the experimental treatment on the concentration of urinary ketones
Impact of plasma glucose modifications on progression free survival | 40 months
  Impact of plasma glucose modifications during the treatment on progression free survival
Impact of serum insulin modifications on progression free survival | 40 months
  Impact of serum insulin modifications during the treatment on progression free survival
Impact of serum IGF-1 modifications on progression free survival | 40 months
  Impact of serum IGF-1 modifications during the treatment on progression free survival
Impact of urinary ketone bodies on progression free survival | 40 months
  Impact of urinary ketone body modifications during the treatment on progression free survival
Impact of lipid profile modifications on progression free survival | 40 months
  Impact of lipid profile modifications during the treatment on progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Marina Chiara Garassino, M.D., Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Marina Chiara Garassino, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ding L, Getz G, Wheeler DA, Mardis ER, McLellan MD, Cibulskis K, Sougnez C, Greulich H, Muzny DM, Morgan MB, Fulton L, Fulton RS, Zhang Q, Wendl MC, Lawrence MS, Larson DE, Chen K, Dooling DJ, Sabo A, Hawes AC, Shen H, Jhangiani SN, Lewis LR, Hall O, Zhu Y, Mathew T, Ren Y, Yao J, Scherer SE, Clerc K, Metcalf GA, Ng B, Milosavljevic A, Gonzalez-Garay ML, Osborne JR, Meyer R, Shi X, Tang Y, Koboldt DC, Lin L, Abbott R, Miner TL, Pohl C, Fewell G, Haipek C, Schmidt H, Dunford-Shore BH, Kraja A, Crosby SD, Sawyer CS, Vickery T, Sander S, Robinson J, Winckler W, Baldwin J, Chirieac LR, Dutt A, Fennell T, Hanna M, Johnson BE, Onofrio RC, Thomas RK, Tonon G, Weir BA, Zhao X, Ziaugra L, Zody MC, Giordano T, Orringer MB, Roth JA, Spitz MR, Wistuba II, Ozenberger B, Good PJ, Chang AC, Beer DG, Watson MA, Ladanyi M, Broderick S, Yoshizawa A, Travis WD, Pao W, Province MA, Weinstock GM, Varmus HE, Gabriel SB, Lander ES, Gibbs RA, Meyerson M, Wilson RK. Somatic mutations affect key pathways in lung adenocarcinoma. Nature. 2008 Oct 23;455(7216):1069-75. doi: 10.1038/nature07423. PMID 18948947
- [Result] Chen Z, Fillmore CM, Hammerman PS, Kim CF, Wong KK. Non-small-cell lung cancers: a heterogeneous set of diseases. Nat Rev Cancer. 2014 Aug;14(8):535-46. doi: 10.1038/nrc3775. PMID 25056707
- [Result] McCleland ML, Adler AS, Deming L, Cosino E, Lee L, Blackwood EM, Solon M, Tao J, Li L, Shames D, Jackson E, Forrest WF, Firestein R. Lactate dehydrogenase B is required for the growth of KRAS-dependent lung adenocarcinomas. Clin Cancer Res. 2013 Feb 15;19(4):773-84. doi: 10.1158/1078-0432.CCR-12-2638. Epub 2012 Dec 6. PMID 23224736
- [Result] Hanahan D, Weinberg RA. Hallmarks of cancer: the next generation. Cell. 2011 Mar 4;144(5):646-74. doi: 10.1016/j.cell.2011.02.013. PMID 21376230
- [Result] Vernieri C, Casola S, Foiani M, Pietrantonio F, de Braud F, Longo V. Targeting Cancer Metabolism: Dietary and Pharmacologic Interventions. Cancer Discov. 2016 Dec;6(12):1315-1333. doi: 10.1158/2159-8290.CD-16-0615. Epub 2016 Nov 21. PMID 27872127
- [Result] Shaw RJ, Bardeesy N, Manning BD, Lopez L, Kosmatka M, DePinho RA, Cantley LC. The LKB1 tumor suppressor negatively regulates mTOR signaling. Cancer Cell. 2004 Jul;6(1):91-9. doi: 10.1016/j.ccr.2004.06.007. PMID 15261145
- [Result] Shaw RJ, Kosmatka M, Bardeesy N, Hurley RL, Witters LA, DePinho RA, Cantley LC. The tumor suppressor LKB1 kinase directly activates AMP-activated kinase and regulates apoptosis in response to energy stress. Proc Natl Acad Sci U S A. 2004 Mar 9;101(10):3329-35. doi: 10.1073/pnas.0308061100. Epub 2004 Feb 25. PMID 14985505
- [Result] Shackelford DB, Shaw RJ. The LKB1-AMPK pathway: metabolism and growth control in tumour suppression. Nat Rev Cancer. 2009 Aug;9(8):563-75. doi: 10.1038/nrc2676. PMID 19629071
- [Result] Zhou G, Myers R, Li Y, Chen Y, Shen X, Fenyk-Melody J, Wu M, Ventre J, Doebber T, Fujii N, Musi N, Hirshman MF, Goodyear LJ, Moller DE. Role of AMP-activated protein kinase in mechanism of metformin action. J Clin Invest. 2001 Oct;108(8):1167-74. doi: 10.1172/JCI13505. PMID 11602624
- [Result] Shackelford DB, Abt E, Gerken L, Vasquez DS, Seki A, Leblanc M, Wei L, Fishbein MC, Czernin J, Mischel PS, Shaw RJ. LKB1 inactivation dictates therapeutic response of non-small cell lung cancer to the metabolism drug phenformin. Cancer Cell. 2013 Feb 11;23(2):143-58. doi: 10.1016/j.ccr.2012.12.008. Epub 2013 Jan 24. PMID 23352126
- [Result] Lee C, Raffaghello L, Brandhorst S, Safdie FM, Bianchi G, Martin-Montalvo A, Pistoia V, Wei M, Hwang S, Merlino A, Emionite L, de Cabo R, Longo VD. Fasting cycles retard growth of tumors and sensitize a range of cancer cell types to chemotherapy. Sci Transl Med. 2012 Mar 7;4(124):124ra27. doi: 10.1126/scitranslmed.3003293. Epub 2012 Feb 8. PMID 22323820
- [Result] Safdie FM, Dorff T, Quinn D, Fontana L, Wei M, Lee C, Cohen P, Longo VD. Fasting and cancer treatment in humans: A case series report. Aging (Albany NY). 2009 Dec 31;1(12):988-1007. doi: 10.18632/aging.100114. PMID 20157582
- [Result] de Groot S, Vreeswijk MP, Welters MJ, Gravesteijn G, Boei JJ, Jochems A, Houtsma D, Putter H, van der Hoeven JJ, Nortier JW, Pijl H, Kroep JR. The effects of short-term fasting on tolerance to (neo) adjuvant chemotherapy in HER2-negative breast cancer patients: a randomized pilot study. BMC Cancer. 2015 Oct 5;15:652. doi: 10.1186/s12885-015-1663-5. PMID 26438237
- [Result] Dorff TB, Groshen S, Garcia A, Shah M, Tsao-Wei D, Pham H, Cheng CW, Brandhorst S, Cohen P, Wei M, Longo V, Quinn DI. Safety and feasibility of fasting in combination with platinum-based chemotherapy. BMC Cancer. 2016 Jun 10;16:360. doi: 10.1186/s12885-016-2370-6. PMID 27282289
- [Result] Wei M, Brandhorst S, Shelehchi M, Mirzaei H, Cheng CW, Budniak J, Groshen S, Mack WJ, Guen E, Di Biase S, Cohen P, Morgan TE, Dorff T, Hong K, Michalsen A, Laviano A, Longo VD. Fasting-mimicking diet and markers/risk factors for aging, diabetes, cancer, and cardiovascular disease. Sci Transl Med. 2017 Feb 15;9(377):eaai8700. doi: 10.1126/scitranslmed.aai8700. PMID 28202779
- [Result] Di Biase S, Lee C, Brandhorst S, Manes B, Buono R, Cheng CW, Cacciottolo M, Martin-Montalvo A, de Cabo R, Wei M, Morgan TE, Longo VD. Fasting-Mimicking Diet Reduces HO-1 to Promote T Cell-Mediated Tumor Cytotoxicity. Cancer Cell. 2016 Jul 11;30(1):136-146. doi: 10.1016/j.ccell.2016.06.005. PMID 27411588